CLINICAL TRIAL: NCT00505349
Title: Blood Neurotrophic Factors in Adults
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Collaborators: University of California, San Francisco (Other); Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OUT-117-2005
Record Dates: First submitted 2007-07-19; First posted 2007-07-23 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Healthy
Keywords: neurotrophic factors; cognitive status; young adults; mature adults; cognitive training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Intervention Arm (No Intervention): Phase I in this study will involve the evaluation of blood-derived neurotrophic factors in healthy, younger adults (18-30.) Individuals in this group will not undergo computerized, cognitive training.
- Cognitive Training (Experimental): Phase II of this study will involve an evaluation of the pre- and post- cognitive training levels of blood-derived neurotrophic factors in healthy, mature adults. Participants randomized to this arm will receive SAAGE-based computerized cognitive training.
  Interventions: Behavioral: Computer-based cognitive training

INTERVENTIONS:
Behavioral: Computer-based cognitive training — The experimental cognitive training program consists of interactive training exercises in which the participant responds to visual patterns and stimuli. The program is designed upon the principles of brain-plasticity, and, for the purposes of this study, is intended to be used for an 8-10 week period (40 total hours of training.)
  Arms: Cognitive Training

SUMMARY:
The overall goal of this study is to evaluate the impact of cognitive training on blood levels of neurotrophic factors in adults.

DETAILED DESCRIPTION:
Current research suggests that levels of brain-derived neurotrophic factor (BDNF) and certain excitatory neurotransmitters - specifically glutamate, D-serine, and glycine are low in participants with depression and other mental illnesses (Wolkowitz and Reus 2002, Tan et al., 2005; Shoval & Weizman, 2005; Hashimoto et al., 2005). Research also suggests that levels of both BDNF and excitatory transmitters can be enhanced by cognitive stimulation (Hynd et al., 2005; Wu et al., 2005; Yang et al., 2005; Mattson et al., 2004). BDNF is found in brain tissue and is also measurable in blood; it stimulates neuronal cell growth in certain brain regions (Duman, 2004). In Phase 1, we wish to measure the levels of specific neurotrophic factors in healthy, young participants. Phase 2 is intended to correlate similar levels with change in neurocognitive performance in healthy, older participants. Overall, this study is designed to obtain a raw measure of the impact that cognitive training has on the mature adult brain.

ELIGIBILITY:
Inclusion Criteria:

Phase 1: Closed

* Age 18-30 at the time of consent
* Good general medical health
* Willing to undergo venipuncture procedure

Phase 2: Activation Pending

* Age 65 or older at the time of consent
* Mini-Mental Status Examination (MMSE) score of 26 or higher
* Willing to undergo venipuncture procedure
* Fluency in the English language
* Participant is willing and able to commit to the time requirement of the study

Exclusion Criteria:

Phase 1

* Participant is experiencing chronic or acute illness
* Current substance abuse, including alcoholism
* Diagnosis of a major psychological disorder
* Current use, or use within the past 3 months of medications specified by protocol
* Participant is unwilling or unable to perform questionnaires as specified in the protocol
* Participant is not capable of giving informed consent or is unable to comprehend and/or follow directions in English
* Participant is enrolled in a concurrent clinical study that could affect the outcome of this study
* Female only: Participant is pregnant

Phase 2

Sensory/Motor Exclusions:

* Reported or observed difficulties with a participant's dominant hand

Psychiatric Exclusions:

* Current diagnosis of a major psychological disorder or a psychiatric hospitalization
* Current substance abuse, including alcoholism

Neurological Exclusions:

* Current diagnosis of a major neurological disorder that may impact cognitive functioning
* History of stroke, traumatic brain injury (leading to loss of consciousness), brain cancer, or invasive neurological procedure within the past year
* Diagnosis of medically uncontrolled seizure disorder

Medication Exclusions:

* Current use, or use within the past 3 months of medications specified within the investigational plan

Additional Exclusions:

* Participant is unwilling or unable to perform assessments and/or evaluations as specified in the protocol
* Participant is not capable of giving informed consent or is unable to comprehend and/or follow directions
* Participant is enrolled in a concurrent clinical study that could affect the outcome of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome of this study will be the evaluation of blood derived neurotrophic factors in both young adults and in mature adults undergoing cognitive training. | Up to 14 weeks post-enrollment

SECONDARY OUTCOMES:
To obtain information on the levels of growth factors in health adults | Required blood draws at three study intervals

CONTACTS AND LOCATIONS:
Overall Officials: Henry Mahncke, PhD, Principal Investigator — Posit Science Corporation
Locations (1):
- Posit Science Corporation, San Francisco, California, United States